CLINICAL TRIAL: NCT01275365
Title: Optimizing Protein Intake in Older Americans With Mobility Limitations
Acronym: OPTIMen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Shalendar Bhasin, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P001321; 7R01AG037547 (NIH)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Mobility Limitation
Keywords: Mobility Limitation; Low Protein Intake; Older Men; Testosterone
MeSH Terms: conditions — Mobility Limitation | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo/Low Protein (No Intervention): Placebo injections weekly; 0.8 g/kg/day protein
- Placebo/High Protein (No Intervention): Placebo injections weekly; 1.3 g/kg/day protein
- Testosterone/Low Protein (Other): Testosterone enanthate 100 mg intramuscularly weekly; 0.8 g/kg/day protein
  Interventions: Drug: Testosterone enanthate
- Testosterone/High Protein (Other): Testosterone enanthate 100 mg intramuscularly weekly; 1.3 g/kg/day protein
  Interventions: Drug: Testosterone enanthate

INTERVENTIONS:
Drug: Testosterone enanthate — Testosterone enanthate 100 mg intramuscularly weekly
  Arms: Testosterone/Low Protein
Drug: Testosterone enanthate — Testosterone enanthate 100 mg intramuscularly weekly
  Arms: Testosterone/High Protein

SUMMARY:
This will be a randomized, placebo-controlled, parallel group, double blind, clinical trial in community dwelling, older men, 65 years of age or older, who have mobility limitation and low protein intake. The study will have a 2 X 2 factorial design, which will allow us to investigate the effects of dietary protein intake and testosterone separately and together.

DETAILED DESCRIPTION:
The recommended dietary allowance (RDA) for protein, set at 0.8 grams/kg/day for adult men and women, has engendered debate and many experts advocate protein intakes substantially above the RDA to help maintain muscle anabolism in older individuals. It is not known whether increasing protein intake in older Americans, whose current intake is below the RDA, increases skeletal muscle mass, muscle performance and physical function.

Our first aim is to determine whether administration of 1.3 g/kg/day of protein, compared to the RDA (0.8 g/kg/day), will result in greater improvements in lean body mass, maximal voluntary muscle strength and power, and self-reported and performance-based measures of physical function in older men. Our second aim is to determine whether the gains in lean body mass, maximal voluntary strength and self-reported and performance-based measures of physical function during testosterone administration are greater with 1.3 g protein than with the RDA in older men on a eucaloric diet.

We will conduct a randomized, placebo-controlled, double-blind trial using a 2 X 2 factorial design. Community dwelling men, 65 years or older, who have self-reported mobility limitation, a daily protein intake of <0.8 g/kg/day and no contraindications for testosterone therapy, will be randomly assigned to one of four groups: placebo injections plus protein 0.8 g/kg/day; placebo injections plus protein 1.3 g/kg/day; testosterone enanthate 100 mg weekly plus protein 0.8 g/kg/day; testosterone enanthate 100 mg weekly plus protein 1.3 g/kg/day. Treatment duration will be 6 months. The primary outcome is change in lean body mass from baseline to 6 months, measured by dual energy X-ray absorptiometry. Secondary outcomes include change in maximal voluntary strength in leg and chest press exercises, leg power, self-reported (physical function domain of SF-36) and performance-based measures of physical function (6-min walking distance and speed, stair climbing power, and load carrying), fatigue, well-being and affectivity balance. Safety measures include urinary calcium excretion, hematocrit, prostate specific antigen (PSA) and prostate examination.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling men 65 years of age or older
2. A score of 3-10 on the short physical performance battery (SPPB)
3. Daily protein intake less than the recommended daily allowance of 0.83 g/kg/day (from 3 24-hour food recalls)
4. Able to give informed consent

Exclusion Criteria:

1. History of prostate or breast cancer
2. American Urological Association [AUA] symptom index score of >19
3. Prostate specific antigen (PSA) >4 ng/ml in White men or >3 ng/ml in Black men
4. Prostate specific antigen (PSA) > 4 ng/ml in non-Black men or >3 ng/ml in Black men. These subjects may be enrolled if they have a negative transrectal biopsy within the past year.
5. Myocardial infarction or stroke within the last 6 months
6. Uncontrolled congestive heart failure, based on the study physician's evaluation
7. Serum creatinine > 2.0 mg/dL; men on any kind of dialysis will be excluded.
8. History of celiac disease, Crohn's disease, or ulcerative colitis
9. History of any malignancy requiring treatment within the previous 2 years, except non-melanic skin cancers. Men with cancers who have not required active treatment within the past two years and who have not had disease recurrence within the past two years may be enrolled at the discretion of the study physician.
10. Neuromuscular diseases: motor neuron diseases, multiple sclerosis, adult muscular dystrophies, and myasthenia gravis
11. History of stroke with residual limb weakness that affected the individual's ability to walk; subjects with history of stroke who do not have residual limb weakness may be enrolled.
12. Schizophrenia, bipolar disorder, or untreated diagnosed depression. Subjects with unipolar depression who are on an antidepressant medication are eligible.
13. TSH levels <0.4 or >5 mlU/L
14. Systolic blood pressure (BP) >160 or diastolic BP >100 mm Hg (average of 2 measurements taken at Visit 1)
15. Hemoglobin A1c >8.0% or taking insulin. Men with diabetes mellitus whose A1C is less than 8.0% or who are not taking insulin will be eligible.
16. Mini-Mental Status Exam [MMSE] <24
17. Body mass index (BMI) less than 20 or greater than 40 kg/m2
18. Not willing to eat all of the following: red meat, eggs, poultry, fish and shellfish
19. Allergy to sesame, peanuts, soy, gluten or shellfish
20. Current alcohol use >21 drinks/week based on self-report
21. Confinement to a wheelchair
22. Use of anabolic therapies (Testosterone, DHEA, androstenedione, rhGH) within the past year
23. Current use of levodopa or anticoagulants
24. Current enrollment in a structured weight management program or participation in any weight intervention studies in the last 90 days
25. Serum ALT and AST greater than 3 x upper limit of normal
26. Hematocrit < 30% or >48%
27. Subject is not able to eat 3 frozen study meals per day for 6 months
28. Subject is unwilling to stop current nutritional supplements
29. Progressive intensive resistance training within 12 weeks of screening
30. Non-compliant with run-in diet and/or supplement

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-05; Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Huang G, Pencina K, Li Z, Apovian CM, Travison TG, Storer TW, Gagliano-Juca T, Basaria S, Bhasin S. Effect of Protein Intake on Visceral Abdominal Fat and Metabolic Biomarkers in Older Men With Functional Limitations: Results From a Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2021 May 22;76(6):1084-1089. doi: 10.1093/gerona/glab007. PMID 33417663
- [Derived] Krok-Schoen JL, Archdeacon Price A, Luo M, Kelly OJ, Taylor CA. Low Dietary Protein Intakes and Associated Dietary Patterns and Functional Limitations in an Aging Population: A NHANES analysis. J Nutr Health Aging. 2019;23(4):338-347. doi: 10.1007/s12603-019-1174-1. PMID 30932132
- [Derived] Bhasin S, Apovian CM, Travison TG, Pencina K, Moore LL, Huang G, Campbell WW, Li Z, Howland AS, Chen R, Knapp PE, Singer MR, Shah M, Secinaro K, Eder RV, Hally K, Schram H, Bearup R, Beleva YM, McCarthy AC, Woodbury E, McKinnon J, Fleck G, Storer TW, Basaria S. Effect of Protein Intake on Lean Body Mass in Functionally Limited Older Men: A Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):530-541. doi: 10.1001/jamainternmed.2018.0008. PMID 29532075
- [Derived] Apovian CM, Singer MR, Campbell WW, Bhasin S, McCarthy AC, Shah M, Basaria S, Moore LL. Development of a Novel Six-Month Nutrition Intervention for a Randomized Trial in Older Men with Mobility Limitations. J Nutr Health Aging. 2017;21(10):1081-1088. doi: 10.1007/s12603-017-0990-4. PMID 29188864

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Started | 24 | 24 | 22 | 22
Completed | 21 | 21 | 17 | 19
Not Completed | 3 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein | Total
Number analyzed (Participants) | 24 | 24 | 22 | 22 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (4.2) | 73.5 (5.7) | 71.0 (3.6) | 76.0 (7.9) | 73.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 24 | 24 | 22 | 22 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 22 | 22 | 92
Body weight [Mean (Standard Deviation); unit: kg] | 95.3 (12.5) | 90.2 (15.8) | 94.4 (17.6) | 87.2 (18.3) | 91.8 (16.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (4.2) | 29.6 (4.6) | 31.4 (5.5) | 29.0 (5.0) | 30.3 (4.9)
Diabetes [Count of Participants; unit: Participants] | 4 | 4 | 3 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry (DXA)
Description: Primary outcome is change in lean body mass, measured by dual energy X-ray absorptiometry (DXA)
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 21 | 21 | 17 | 19
kg | 0.14 (0.31) | 0.74 (0.33) | 4.43 (0.48) | 4.13 (0.42)

2. Secondary Outcome: Change of Maximal Voluntary Strength
Description: Tests of Muscle Performance: (1) Maximal voluntary strength measured by 1-repetition maximum method in leg press; (2) Maximal voluntary strength in chest press; this exercise was chosen because it involves the large muscle groups of the upper extremities.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: newton
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 13 | 9 | 14 | 13
newton
  Maximal voluntary strength in leg press | 134.6 (46.4) | 156.0 (89.1) | 201.8 (44.4) | 191.4 (38.0)
  Maximal voluntary strength in chest press | 41.5 (12.3) | 16.6 (9.2) | 64.5 (11.9) | 59.3 (11.3)

3. Secondary Outcome: Change of Leg Press Power
Description: Muscle Performance measured using Power of hip and knee extension by Bassey's leg rig.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: watts
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 12 | 9 | 15 | 12
watts | 26.9 (17.0) | 96.9 (19.6) | 61.5 (22.2) | 81.7 (16.1)

4. Secondary Outcome: Change of 6-minute Walking Distance
Description: Tests of Physical Function and Task-Specific Performance measured by 6-min walking distance
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 16 | 14 | 16 | 18
meters | 44.2 (17.9) | 49.9 (14.2) | 38.2 (21.9) | 25.5 (11.5)

5. Secondary Outcome: Change of Stair Climbing Tests
Description: Tests of Physical Function and Task-Specific Performance measured by Stair-climbing power +/- 20% load carry. Physical Function was evaluated using two tests of stair climb power using an indoor 12-step staircase. One test consisted of ascending the 12-steps as rapidly as possible without running (unloaded stair climb) while the second test required participants to carry a load equivalent to 20% of their baseline body weight evenly distributed in two canvas tote bags (loaded stair climb). Time to ascend the stairs was measured electronically with a digital clock and switch mats placed at the base of the steps and on the 12th step. Power in watts is calculated by the following: [body weight (kilograms) * distance (meters)/ (time/60)] /6.12.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: watts
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 14 | 11 | 16 | 15
watts
  Unloaded | 50.8 (19.2) | 55.4 (14.2) | 53.2 (17.5) | 4.2 (13.5)
  Loaded | 56.8 (15.7) | 83.7 (28.5) | 56.6 (18.8) | 26.9 (14.3)

6. Secondary Outcome: Change of 50-meter Loaded Walking Test
Description: Tests of Physical Function and Task-Specific Performance measured by 50-meter timed walk + 20% load carry. Physical Function was evaluated using test of 50-meter loaded walking speed. The test required participants to carry a load equivalent to 20% of their baseline body weight evenly distributed in two canvas tote bags. Time was measured electronically with a digital clock. Speed in meters per second is calculated by the following: 50/time.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 11 | 13 | 15 | 13
meters per second | 0.15 (0.04) | 0.11 (0.05) | 0.06 (0.05) | 0.08 (0.04)

7. Secondary Outcome: Change of Self-reported Physical Function Domain of Short Form Health Survey (SF-36)
Description: 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. Physical function domain of the Medical Outcomes Study Short Form-36 (SF-36) contains 10 items with the score range of 0-100. Higher score yields better performance.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 21 | 21 | 17 | 19
units on a scale | -1.4 (3.1) | -5.5 (5.3) | 2.1 (2.8) | -2.9 (2.9)

8. Secondary Outcome: Change of Psychological Well Being Index (PGWBI)
Description: The PGWBI is a 22-item health-related Quality of Life (HRQoL) questionnaire developed in US which produces a self-perceived evaluation of psychological well-being expressed by a summary score. The 22 items are grouped in 6 dimensions. A global score is computed as the sum of all items with range of 0-110. A higher score yields better performance.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 21 | 21 | 17 | 19
units on a scale | -0.56 (1.53) | 1.17 (1.77) | 0.32 (2.08) | 2.68 (1.58)

9. Secondary Outcome: Change of Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale
Description: The FACIT Fatigue Scale is a 13-item questionnaire that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point scale (4 = not at all fatigued to 0 = very much fatigued). Score ranges 0-52. The higher the score, the better the quality of life.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 21 | 21 | 17 | 19
units on a scale | 0.14 (1.56) | -0.14 (1.41) | -0.53 (1.39) | 1.05 (1.16)

10. Secondary Outcome: Change of Derogatis Affective Balance Scale (DABS)
Description: The Derogatis Affects Balance Scale (DABS) is a multidimensional self-report mood and affects inventory comprised of 40 adjective-items using a 5-point Likert style scale. The DABS global scores consist of the Positive Total score (PTOT), Negative Total score (NTOT), where The Positive Affects Total (PTOT) is defined as the sum of all scores on the four positive affects dimensions of joy, contentment, vigor and affection, ranging 0-80. Similarly, the Negative Affects Total (NTOT) is represented as the sum of scores on the four negative dimensions of anxiety, depression, guilt and hostility, ranging 0-80. The Affects Expressiveness Index (AEI) is defined as the sum total of PTOT and NTOT, ranging 0-160. Higher score yields stronger affective intensity.
Time Frame: 6 months from baseline
Population: All randomized and treated participants with data available at the given time-point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
Number analyzed (Participants) | 21 | 20 | 17 | 19
units on a scale
  Affects Expressiveness Index (AEI) | 0.65 (3.54) | 1.45 (1.96) | -0.50 (2.51) | -3.17 (1.99)
  Positive Total score (PTOT) | 1.38 (2.09) | 2.10 (1.70) | 0.69 (1.68) | 1.89 (1.29)
  Negative Total score (NTOT) | -1.50 (2.03) | -0.65 (1.36) | -0.88 (2.85) | -5.53 (1.47)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo/Low Protein | Placebo/High Protein | Testosterone/Low Protein | Testosterone/High Protein
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/24 | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 20/24 | 21/24 | 21/22 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Low Protein (N=24) | Placebo/High Protein (N=24) | Testosterone/Low Protein (N=22) | Testosterone/High Protein (N=22)
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Low Protein (N=24) | Placebo/High Protein (N=24) | Testosterone/Low Protein (N=22) | Testosterone/High Protein (N=22)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pulmonary congestion (Cardiac disorders) | 0 | 2 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear infection (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 2 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 4 (5)
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 (4)
Flatulence, bloating and distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1
Asthma (Immune system disorders) | 1 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 0
Pheumonia (Infections and infestations) | 1 | 2 | 0 | 0
Urinary tract infections (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Epicodylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 | 1 | 1
Injection site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (2) | 0
Biopsy skin (Investigations) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Prostatic specific antigen abnormal (Investigations) | 2 | 2 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Oedema peripheral (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 4 | 3
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 | 2 | 1 (2)
Muscle strain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 (2) | 1 | 3
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 3 (6)
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Gait disturbance (Nervous system disorders) | 0 | 0 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 2 | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 2 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 1 | 4
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatic asymmetry (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0 | 0 | 1
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Ifluenza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 (2) | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Skin ulcer (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT01275365/Prot_SAP_000.pdf